CLINICAL TRIAL: NCT06222619
Title: Effect of Portal Vein Embolization on Surgical Outcomes and Long-term Survival in Patients With Perihilar Cholangiocarcinoma
Brief Title: Effect of PVE on Surgical Outcomes and Long-term Survival in Perihilar Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Other Study IDs: H-2001-092-1095
Record Dates: First submitted 2024-01-11; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Biliary Tract Cancer; Portal Vein Embolization
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Resection without PVE: Resection of bile duct and associated hemi-liver without portal vein embilzation
- Resection after PVE: Resection of bile duct and associated hemi-liver after portal vein embilzation
  Interventions: Procedure: Potal vein embilization
- No resection after PVE: No resection of bile duct and associated hemi-liver after portal vein embilzation
  Interventions: Procedure: Potal vein embilization

INTERVENTIONS:
Procedure: Potal vein embilization — Portal vein of involved bile duct is embolized to increase the volume of remnant liver.
  Other Names: Surgical resection
  Groups: No resection after PVE; Resection after PVE

SUMMARY:
Portal vein embolization is often recommended to reduce the risk of postoperative liver failure and mortality. In this retrospective cohort study, researchers investigated the effect of portal vein embolization in patients with resectable perihilar cholangiocarcinoma bismuth type III and IV.

ELIGIBILITY:
Inclusion Criteria:

1. patients with Bismuth type III or IV stricture on radiological examination, including computed tomography (CT) or magnetic resonance cholangiography
2. patients with perihilar cholangiocarcinoma histologically confirmed by surgical resection or forceps biopsy/brush cytology under endoscopic retrograde cholangiopancreatography or through the percutaneous transhepatic biliary drainage tract.

Exclusion Criteria:

1. patients with unresectable perihilar cholangiocarcinoma
2. patients who refused treatment
3. patients with other concomitant malignancies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Bismuth type III-IV perihilar cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | The time from diagnosis until the date of death or last date of follow-up or end of study up to 24 months
  Overall survival of each group (A-C).

SECONDARY OUTCOMES:
Recurrence free survival | The time from surgical resection until the date of recurrence or death or last date of follow-up or end of study up to 24 months
  Recurrence free survival of patients who underwent surgical resection

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea